CLINICAL TRIAL: NCT03285854
Title: Assessing Calcium Balance in Children With Chronic Kidney Disease to Optimise Treatment Strategies
Brief Title: Calcium Balance Studies in Children With CKD and on Dialysis
Acronym: Cal-Bal
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: University of Kiel (Other); Athens General Children's Hospital "Pan. & Aglaia Kyriakou" (Other); Cukurova University (Other)
Responsible Party: Sponsor
Other Study IDs: 15HM36
Record Dates: First submitted 2017-09-12; First posted 2017-09-18 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Chronic Kidney Disease Mineral and Bone Disorder
Keywords: CKD; Dialysis; calcium; mineral and bone disorder (MBD); calcification; DXA; peripheral quantitative CT scan (pqCT)
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder; Calcinosis; Bone Diseases | interventions — Urination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, urine, stool and dialysis fluid samples will be collected
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with CKD stage 3-5 and dialysis: Children of all ages with an eGFR <60ml/min/1.73m2, including those on dialysis
  Interventions: Diagnostic Test: Collection of blood, urine and stool samples
- Healthy age and gender matched children: 1. All children <18 years
  2. Normal renal function (eGFR 90-120ml/min/1.73m2 [calculated by Schwartz formula] in children >1 year and serum creatinine <35μMol/L in children <1 year)
  3. Weight, height and BMI within 2 SD of normal using WHO growth charts In order to make this study as 'real-life' as possible, free-living UK children on their usual diet and dietary supplementation (including Ca and Vit D), if any, will be included, but analysis will account for medication doses and blood levels.
  Interventions: Diagnostic Test: Collection of blood, urine and stool samples

INTERVENTIONS:
Diagnostic Test: Collection of blood, urine and stool samples — Collection of blood, urine and stool samples, diet diary and bone scans
  Other Names: DEXA - lumbar spine and hips; tibial peripheral quantitative CT; Dietary record

SUMMARY:
This is a novel, non-invasive method of assessing Ca balance by natural Ca isotope fractionation.

DETAILED DESCRIPTION:
Detailed description and study protocol will be available to individuals on request.

ELIGIBILITY:
I - For healthy children

Inclusion criteria

* All children <18 years
* Normal renal function (eGFR 90-120ml/min/1.73m2 [calculated by Schwartz formula] in children >1 year and serum creatinine <35μMol/L in children <1 year)
* Weight, height and BMI within 2 SD of normal using WHO growth charts In order to make this study as 'real-life' as possible, free-living UK children on their usual diet and dietary supplementation (including Ca and Vit D), if any, will be included, but analysis will account for medication doses and blood levels.

Exclusion criteria

* Pre-existing bone disease - inherited or acquired
* Fractures in the preceding 6 months
* Glucocorticoid therapy in the preceding year, or a lifetime cumulative steroid exposure ≥6 months
* Bisphosphonate therapy at any time in the past
* Any acute illness in the preceding 2 weeks (when the child is unable to maintain their usual diet or has bed rest)

II - For CKD and dialysis children

Inclusion criteria

* Children of all ages with an eGFR <60ml/min/1.73m2, including those on dialysis.

Exclusion criteria

* As listed above for healthy children.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All children with chronic kidney disease stage 3-5 and on dialysis and age matched controls
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Calcium isotope fractionation in blood, urine and stool in healthy children and those with CKD | 24 months
  available on request
number of children with fractures, and clinical and biochemical correlates of fractures | 12 months
  available on request
Bone scans - whole body & lumbar spine DEXA, bone mineral density on tibial peripheral quantitative CT scan | 24 months
  available on request

CONTACTS AND LOCATIONS:
Overall Officials: Rukshana C Shroff, MD PhD, Principal Investigator — Great Ormond Street Hospital for Children NHS Foundation Trust
Locations (1):
- Great Ormond Street Hospital for Children NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing will be considered at the end of the study.